CLINICAL TRIAL: NCT03823963
Title: A Monocentric, Comparative and Randomized Study on Pressure Ulcers Prevention With Mepilex® Border Sacrum Dressing in Scheduled Cardiovascular Surgery
Brief Title: Study on Pressure Ulcers Prevention With Mepilex® Border Sacrum Dressing in Scheduled Cardiovascular Surgery
Acronym: MEPICARD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHU-418; 2018-A00694-51 (Other: 2018-A00694-51)
Record Dates: First submitted 2019-01-11; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Pressure Ulcers; Prevention; Skin Ulcer; Ulcer
MeSH Terms: conditions — Pressure Ulcer; Skin Ulcer; Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Other): pressure ulcer prevention standard care
  Interventions: Other: Standard care
- standard care + Mepilex® Border (Experimental): pressure ulcer prevention standard care + Mepilex® Border applied on sacrum
  Interventions: Combination Product: Mepilex® Border dressing; Other: Standard care

INTERVENTIONS:
Combination Product: Mepilex® Border dressing — Soft silicone self-adherent dressing (5-layers)
  Arms: standard care + Mepilex® Border
Other: Standard care — The control group will receive pressure ulcer prevention standard care

SUMMARY:
The study is a randomised controlled trial of patients admitted for a scheduled cardiac surgery at the Clermont-Ferrand hospital.

Patients meeting the study inclusion criteria will be allocated to either the control group that will receive pressure ulcer prevention standard care or the intervention group that will receive pressure ulcer prevention standard care plus have a Mepilex® Border dressing applied to their sacrum.

DETAILED DESCRIPTION:
The main objective of this research is to evaluate the impact of Mepilex Border® dressing applied in addition to standard pressure ulcer prevention protocol, in a French hospital setting, in at-risk patients in a cardiovascular surgery unit with full hospitalisation including block operation and ICU.

Hypothesis: Patients treated with Mepilex® Border dressings will have a lower incidence rate of sacral pressure ulcer development than patients receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years of age,
* Subject programmed to benefit from cardiac surgery with sternotomy,
* Subject capable and willing to comply with the protocol and willing to give his written consent,
* Subject affiliated to a social security system

Exclusion Criteria:

* Subject with a skin lesion in the sacral area upon admission,
* Subject admitted for emergency cardiovascular surgery (unscheduled subject),
* Subject admitted for heart transplant surgery,
* Subject participating in another clinical study or in a period of exclusion from a study previous,
* Subject with a linguistic or psychological disability to sign informed consent,
* Subject refusing to give written consent,
* Subject deprived of liberty by administrative or judicial decision, under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Pressure ulcer incidence | 0-20 days
  Incidence of sacral pressure ulcers acquired during patients' hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Franck HENTZ, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France